CLINICAL TRIAL: NCT05254665
Title: An Open, Multi-cohort, Phase II Clinical Study Evaluating the Efficacy and Safety of Docetaxel Polymer Micelles for Injection in Patients With Advanced Malignant Solid Tumors
Brief Title: A Study of Docetaxel Polymeric Micelles for Injection in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B02B00903-DTAX-201
Record Dates: First submitted 2022-01-19; First posted 2022-02-24 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Docetaxel Polymeric Micelles for Injection (Experimental): Docetaxel Polymeric Micelles for Injection
  Interventions: Drug: Docetaxel Polymeric Micelles for Injection

INTERVENTIONS:
Drug: Docetaxel Polymeric Micelles for Injection — Docetaxel polymeric micelles，usage and quantity of Docetaxel polymeric micelles follows the clinical study proctol，not published.

SUMMARY:
This study is an open, multi-cohort phase II clinical trial, the overall design is divided into two parts: dose confirmation stage and expansion stage. Dose confirmation stage is to evaluate the safety and tolerability of three dosing regimenes of docetaxel polymer micelle for injection in patients with advanced esophageal cancer, and to determine the best dosing regimenes for entering the expansion stage. The expansion stage iwas used to evaluate the efficacy and further safety of the best dosing regimen identified in the dose confirmation stage in patients with advanced solid tumors. All subjects in the dose confirmation stage and expansion stage will continue treatment according to the injection docetaxel micelle regimen they received at enrollment until the disease progresses or the investigator determines that continuing treatment with the study drug will not benefit, or any intolerable toxicity occurs, or they voluntarily withdraw, or for other reasons, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female aged 18~75 years old
* Patients with histopathologically or cytologically confirmed advanced or metastatic solid tumors who have failed or are not eligible for standard therapy in the past
* Have an Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* There are measurable tumors(RECIST 1.1)

Exclusion Criteria:

* Previous palliative chemotherapy with docetaxel failed
* Central nervous system metastasis or meningeal metastasis with clinical symptoms
* Has a history of serious cardiovascular disease
* A history of immunodeficiency, including a positive test for human immunodeficiency virus (HIV)
* Active hepatitis B (HBsAg positive, HBV DNA>; ULN) or hepatitis C (HCV antibody positive and HCV RNA>ULN)
* Has a history of allergies to yew medications
* Pregnant or lactating women
* The investigator considered that there were other reasons for the subjects' ineligibility for this clinical study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2022-02 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Dose confirmation stage: Safety and tolerability to determine the subsequent recommended dosing regimen | 2 years
  Incidence of DLT（Dose limited toxicity）
Expansion stage: effect，ORR(Objective Response Rate ) by investigator | 2 years
  Proportion of subjects who have a complete or partial response relative to baseline as assessed by investigator according to RECIST 1.1 criteria

SECONDARY OUTCOMES:
Dose confirmation stage: Objective Response Rate（ORR） by investigator | 2 years
  Proportion of subjects who have a complete or partial response relative to baseline as assessed by investigator according to RECIST 1.1 criteria
Dose confirmation stage: Objective Response Rate（DoR）by investigator | 2 years
  Measured from the date of partial or complete response to therapy until the cancer progresses based on RECIST v1.1 criteria
Dose confirmation stage: Progression free survival（PFS） by investigator | 2 years
  PFS was defined as the time from the date of randomization to the first documented disease progression or death, whichever occurred first. Progression was based on tumor assessment according to the RECIST 1.1 criteria
Dose confirmation stage: Disease Control Rate（DCR）by investigator | 2 years
  Proportion of subjects who have a complete or partial response, or stable disease relative to baseline as assessed by investigator according to RECIST 1.1 criteria
Dose confirmation stage: Overall Survival（OS）by investigator | 2 years
  OS is the time interval from the date of randomization to death from any cause.
Dose confirmation stage: Area under the plasma concentration versus time curve（AUC） | Day 1 to Day 3 of Cycle 1，each cycle is 21 （queue A and C）or 28 days（queue B）
  Area under the plasma concentration versus time curve
Dose confirmation stage: Peak Plasma Concentration（Cmax） | Day 1 to Day 3 of Cycle 1，each cycle is 21 （queue A and C）or 28 days（queue B）
  Peak Plasma Concentration，Maximum concentration of HT001 derived from plasma concentration-time profile
Dose confirmation stage: Time to Peak（Tmax） | Day 1 to Day 3 of Cycle 1，each cycle is 21 （queue A and C）or 28 days（queue B）
  Time of peak blood concentration of HT001 derived from plasma concentration-time profile
Dose confirmation stage: Half-life（t1/2） | Day 1 to Day 3 of Cycle 1，each cycle is 21 （queue A and C）or 28 days（queue B）
  Half-life of HT001 derived from plasma concentration-time profile
Dose confirmation stage: Clearance（CL） | Day 1 to Day 3 of Cycle 1，each cycle is 21 （queue A and C）or 28 days（queue B）
  Clearance of HT001 derived from plasma concentration-time profile
Dose confirmation stage: Volume of distribution（Vd） | Day 1 to Day 3 of Cycle 1，each cycle is 21 （queue A and C）or 28 days（queue B）
  Volume of distribution of HT001 derived from plasma concentration-time profile
Dose confirmation stage: Mean Residence Time（MRT） | Day 1 to Day 3 of Cycle 1，each cycle is 21 （queue A and C）or 28 days（queue B）
  Mean Residence Time of HT001 derived from plasma concentration-time profile
Expansion stage: Objective Response Rate（DoR）by investigator | 2 years
  Measured from the date of partial or complete response to therapy until the cancer progresses based on RECIST v1.1 criteria
Expansion stage：Progression free survival（PFS） by investigator | 2 years
  PFS was defined as the time from the date of randomization to the first documented disease progression or death, whichever occurred first. Progression was based on tumor assessment according to the RECIST 1.1 criteria
Expansion stage：Disease Control Rate（DCR）by investigator | 1.5 year
  Proportion of subjects who have a complete or partial response, or stable disease relative to baseline as assessed by investigator according to RECIST 1.1 criteria
Expansion stage：Overall Survival（OS）by investigator | 2 years
  OS is the time interval from the date of randomization to death from any cause.
Expansion stage: The incidence and severity of adverse events (AEs) and serious adverse events (SAEs) | 2 years
  Frequency and severity of Adverse Events or Serious Adverse Events as defined by CTCAE version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Ye Guo, Ph.D, Principal Investigator — Shanghai East Hospital
Locations (10):
- China (10):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - The Forth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - Shandong Cancer Hospital, Jinan, Shandong
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Tianjin Medical University Cancer Institute&Hospital, Tianjin, Tianjin Municipality
  - Jinhua Municipal Hospital Medical Group, Jinhua, Zhejiang

IPD SHARING:
Plan to Share IPD: No